CLINICAL TRIAL: NCT05649228
Title: A Double-Blind, Randomized, Pilot Study to Investigate the Thermosensitivity of a Topical Palmitated Formulation of Capsaicin
Brief Title: Thermosensitivity of a Topical Palmitated Formulation of Capsaicin
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Chorda Pharma, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-21-1214
Record Dates: First submitted 2022-11-30; First posted 2022-12-14 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Capsaicin

STUDY DESIGN:
Intervention Model Description: Each subject will be given two of either:
  1. vehicle cream containing 0.25% capsaicin palmitate
  2. vehicle cream containing 0.10% non-palmitated capsaicin
  3. vehicle cream alone (placebo)
Who Masked: Participant, Investigator
Masking Description: Labeling codes will be used for a double-blind procedure. Packaging is done by Chorda Pharma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Capsaicin Palmitate (Experimental): Cream containing 0.25% capsaicin palmitate will be applied to an 8 cm2 area of skin on the subject's forearm
  Interventions: Drug: Capsaicin 0.1% Cream; Drug: Placebo Cream
- Capsaicin (Active Comparator): Cream containing 0.1% capsaicin will be applied to an 8 cm2 area of skin on the subject's forearm
  Interventions: Drug: Capsaicin Palmitate 0.25% Cream; Drug: Placebo Cream
- Placebo Cream (Placebo Comparator): Placebo cream will be applied to an 8 cm2 area of skin on the subject's forearm
  Interventions: Drug: Capsaicin 0.1% Cream; Drug: Capsaicin Palmitate 0.25% Cream

INTERVENTIONS:
Drug: Capsaicin 0.1% Cream — A small amount of cream about the size of a U.S. quarter containing 0.10% non-palmitated capsaicin will be applied to participant's forearm using gloved fingers with visible cream left on the surface for one hour.
  Other Names: Zostrix
  Arms: Capsaicin Palmitate; Placebo Cream
Drug: Capsaicin Palmitate 0.25% Cream — A small amount of cream about the size of a U.S. quarter containing 0.25% capsaicin palmitate will be applied to participant's forearm using gloved fingers with visible cream left on the surface for one hour.
  Other Names: Capsadyn
  Arms: Capsaicin; Placebo Cream
Drug: Placebo Cream — A small amount of cream about the size of a U.S. quarter will be applied to participant's forearm using gloved fingers with visible cream left on the surface for one hour.
  Arms: Capsaicin; Capsaicin Palmitate

SUMMARY:
This is a study of the effects of capsaicin, the ingredient that makes hot peppers hot. Capsaicin is currently used in topical ointments to provide temporary relief of minor aches and joint pain associated with arthritis, simple backache, strains, and sprains.

This is a pilot research study that compares the potential of two different capsaicin creams to cause irritation or burning sensation when a small amount (about the size of a quarter) is applied to each forearm of a participant. The amount of capsaicin used in the creams is the same as those found in over-the-counter capsaicin products. The test creams are experimental.

DETAILED DESCRIPTION:
The study design will detect levels of patient dysesthesia in response to Capsadyn using a three-arm, group comparison. Capsadyn will be compared to an active control [capsaicin alone (Cap)], and to a placebo cream alone (PL). The design will use a double-blind for assignment of test article to the three arms. Both the test article administrator and patient will be blinded to test article identity. The test article will be packaged in a coded, white-label, jar with cotton swab applicator.

Participants. Participants for the clinical trial will be recruited through the Carilion Clinic Dermatology Department in Roanoke, VA. In order to minimize the skin area exposed to capsaicin, test articles will be administered to about an 8 cm2 area of the volar forearm. Subject will be informed of the possibility of a transient capsaicin-induced burning sensation along with redness.

Study Groups. The groups are designated Pal and Cap or PL, a placebo (PL) group. The capsaicin drugs are topical analgesics for the temporary relief of minor aches and pains of muscles and joints associated with arthritis. Pal is 0.25% palmitated capsaicin. Cap is 0.10% capsaicin alone and is an active comparator. PL is vehicle alone. Test articles will be balanced arm-to-arm by Pal/Cap, Pal/PL, Cap/PL. Pretest baseline scores will be compared to treatment scores by one-way ANOVA followed by post-hoc analyses for Pal vs PL, Pal vs Cap, and Cap vs PL.

An active comparator is used since non-palmitated capsaicin (unprotected) produces heat. The sensory stimuli would break a neutral control such as vehicle alone. Zostrix at 0.1% capsaicin was used as the active comparator (Cap), a commercially-available topical capsaicin analgesic sold over-the-counter. The concentration of 0.25% capsaicin for Capsadyn (Pal), was based on the upper-limit concentration for capsaicin as specified by the FDA Tentative Final Monograph. A PL group is included since the placebo effect has to be assumed to be intrinsic to pharmaceutical intervention studies. If a placebo effect occurs that would interfere with assessment of the test article intervention, then those assessments can be evaluated with respect to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* 35 to 75 years of age
* Has two arms
* Has intact, unscarred skin over forearms
* Absence of any eczema, hyperkeratosis, scleroderma or other dermatological conditions afflicting the area of test article application that may interfere with absorption as determined by the PI.
* Must agree to not wash forearms during the study period unless a highly uncomfortable burning sensitivity occurs.
* Must be willing to use treatments blinded.
* Must be willing and able to comply with protocol requirements for the duration of study participation, including answering VAS queries in good faith and as diligently as possible.

Exclusion Criteria:

* Younger than 35 and older than 75 years of age
* No previous use of capsaicin products for 48 hours prior to time 0 (application) of test articles.
* Any dermatological conditions that in the judgement of the study site investigator has the potential to disrupt skin integrity or alter sensory function on the forearms.
* Any skin infection, skin irritation (e.g. poison oak), history of eczema, trauma or burn (including sunburn) on the forearms within 30 days preceding application of test article.
* Any recent medical history of painful conditions, surgery, or injury involving or affecting the forearms that may impede skin sensitivity.
* Use of any topically applied products at any location, including prescription or over-the-counter (OTC) analgesic creams/lotions/patches, non-steroidal anti-inflammatory drugs, counter-irritants, local anesthetics, steroids 24 hours prior to the application visit.
* History or current substance abuse including alcoholism/alcohol abuse, as judged by the study site investigator.
* History of hypersensitivity to capsaicin (i.e. chili peppers or OTC capsaicin products).
* At least 30 days since prior topical medications to the skin of the forearms except for emollients or sunscreens.
* No concurrent therapy that may interfere with clinical evaluations.
* No concurrent enrollment in another clinical trial.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Determine any change in relative burning potential for capsaicin palmitate in comparison to non-palmitated capsaicin and to placebo. | Assess for changes every 10 minutes after application for one hour
  Subject assessment of any changes in the presence of a burn using a VAS scale 0 to 10 for both areas of the forearms where topical cream was applied.

SECONDARY OUTCOMES:
Determine the presence and time course of erythema. | Assessed every 10 minutes after application for one hour
  The presence of erythema will be noted and qualified by a clinician erythema assessment scale of 1-4 with 1 being almost clear of redness and 4 being severe redness.
Determine the presence and time course of skin irritation | Assessed every 10 minutes after application for one hour
  Subjects will be asked to assess any tingling, burning, soothing, freezing, and itching of the skin in the area where the topical cream was applied.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Holcomb, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Data will be made available to investigative parties in publication format after study analysis is complete which will include de-identified participant data.

DOCUMENTS (1):
  • Informed Consent Form (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT05649228/ICF_000.pdf